CLINICAL TRIAL: NCT03935802
Title: Analysis of Circulating Epithelial Tumor Cells in Peripheral Blood in Patients With Primary Non-metastatic Breast Cancer Under Adjuvant Radiotherapy
Status: Completed | Type: Observational
Sponsor: University of Jena (Other)
Responsible Party: Principal Investigator, Matthias Mäurer, Dr. Matthias Mäurer, University of Jena
Other Study IDs: CETC 001
Record Dates: First submitted 2019-04-24; First posted 2019-05-02 (Actual); Last update posted 2019-05-02 (Actual); Status verified 2019-04

CONDITIONS: Breast Cancer Female
Keywords: Radiotherapy; CETC; CTC; breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Radiation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- primary non-metastatic breast cancer: primary non-metastatic breast cancer
  Interventions: Radiation: radiation

INTERVENTIONS:
Radiation: radiation

SUMMARY:
The aim of this study was to investigate the systemic effect of radiotherapy on patients with primary non-metastatic breast cancer using CETC and to analyze possible changes in CETC quantity under adjuvant radiotherapy.

DETAILED DESCRIPTION:
In cooperation with the Women's Hospital of the Friedrich Schiller University in Jena, a total of 161 patients with clinically proven, primarily non-metastatic breast cancer were sampled and examined before and after radiotherapy over a period from 09/2002 to 09/2012. The MAINTRAC method was used to quantitatively determine the amount of CETC in the blood and to observe its peritherapeutic course.

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed invasive breast carcinoma
* age >= 18 years
* exclusive treatment at the Jena University Hospital
* complete curative-intended adjuvant or definite radiotherapy
* at least 2 blood collections (before the start of therapy, after the end of the RT)

Exclusion Criteria:

* presence of metastases
* recurrence
* DCIS, inflammatory breast cancer
* second malignancy <10 years before diagnosis of breast cancer
* radiotherapeutic pretreatment

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Primary non-metastatic breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 161 (Actual)
Dates: Start 2002-09-01 (Actual); Primary Completion 2012-09-01 (Actual); Study Completion 2018-09-01 (Actual)

PRIMARY OUTCOMES:
Overall survival | up to 10 years
  from the start of Radiotherapy until death / last seen during follow up

SECONDARY OUTCOMES:
Disease free survival | up to 10 years
  from the start of Radiotherapy until relapse or metastasis / last seen during follow up

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Radiooncology, Jena, Jena, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Maurer M, Schott D, Pizon M, Drozdz S, Wendt T, Wittig A, Pachmann K. Increased Circulating Epithelial Tumor Cells (CETC/CTC) over the Course of Adjuvant Radiotherapy Is a Predictor of Less Favorable Outcome in Patients with Early-Stage Breast Cancer. Curr Oncol. 2022 Dec 24;30(1):261-273. doi: 10.3390/curroncol30010021. PMID 36661670